CLINICAL TRIAL: NCT04781296
Title: Spectral Computed Tomography With Photon-counting Detector
Brief Title: Spectral CT With Advanced CT Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Collaborators: Prismatic Sensors AB (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 20201218-01
Record Dates: First submitted 2021-02-18; First posted 2021-03-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: CT Photon-Counting

STUDY DESIGN:
Intervention Model Description: The single group model will enroll subjects from 5 anatomical areas (lungs, brain/carotid vessels, heart/chest, MSK and abdomen) where CT imaging is applicable and where data on the photon-counting CT is needed to assess feasibility and guide further development of the technology.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Subject's Scanned with Investigational Device (Experimental)
  Interventions: Device: CT with a photon-counting detector

INTERVENTIONS:
Device: CT with a photon-counting detector — Enrolled subjects will complete an exam using the photon-counting CT, with or without IV contract as indicated. Images will then be compared with the previously acquired CT conducted as standard of care.

SUMMARY:
The purpose of the study is to collect data to evaluate feasibility of the using photon-counting CT in a clinical setting.

DETAILED DESCRIPTION:
Data collected in this study includes an assessment of image quality parameters including spatial resolution, image contrast, and noise that will evaluate the product and how this photon-counting CT technology can be used to reduce the overall radiation dose in CT imaging, and enhance clinical applications for CT technology.

ELIGIBILITY:
Inclusion Criteria:

* Age >50 years
* Male
* Normal renal function per standardized guidelines (GFR > 60 mL/min)
* Previous CT examination at KS no more than 12 months prior to the study examination
* Signed informed consent

Exclusion Criteria:

* Iodine contrast is contraindicated.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
Evaluate feasibility of the photon-counting CT in a clinical setting. | 1 year
  The primary objective of this study is to collect and evaluate raw CT scan data collected using the photon-counting CT.

SECONDARY OUTCOMES:
Collect feedback on performance and images generated on the photon-counting CT. | 1 year
  Gather feedback on the performance and image quality of the reconstructed images produced by using the photon-counting CT.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Challman, Study Director — GE Healthcare
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No